CLINICAL TRIAL: NCT06080009
Title: Analysis of Molecular Biomarkers in Periocular Adnexal Tumours
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Savino Gustavo, Professor, Director of Ocular Oncology Unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5896
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Sebaceous Cell Tumor of Eyelid
MeSH Terms: interventions — Exome Sequencing; Retrospective Studies; Exome; Longitudinal Studies

STUDY DESIGN:
Intervention Model Description: Single-centre interventional study on biological sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with Ca sebaceous of the ocular adnexa. (Experimental): adult patients diagnosed with Ca sebaceous of the ocular adnexa.
  Interventions: Genetic: exome sequencing (retrospective) and exome and methylome sequencing (prospective)

INTERVENTIONS:
Genetic: exome sequencing (retrospective) and exome and methylome sequencing (prospective) — Three to nine sections will be used as the source of DNA for each tumor. The pathologist will identify and separate tumor tissue from normal tissue, and the two DNAs will be sequenced separately. Variants obtained from tumor and normal tissue will be compared, with different outcomes. Expected in this way are 1) somatic/tumor-specific variants (which are absent in normal tissue), 2) variants lost during tumor evolution due to segmental chromosomal deletion or other mechanisms that cause loss of heterozygosity. Using these two classes of variants, a clustering analysis will be performed at the end of the sequencing project to better define the phenotype and molecular "signature" of the tumors. In the prospective part of the project, the new tumors will be frozen fresh. This resource will allow methyloma analysis to be performed.

SUMMARY:
The aim of this study is to collect sebaceous carcinomas from the Fondazione Policlinico Gemelli retrospectively and prospectively, to analyse them morphologically and immunopathologically and to correlate them with molecular genetic aspects. This study will help to clarify and develop a more effective multidisciplinary diagnostic-therapeutic pathway.

DETAILED DESCRIPTION:
The purpose of this research is to prospectively and retrospectively collect sebaceous carcinomas from the Fondazione Policlinico Gemelli, examine them immunopathologically and morphologically, and establish a correlation between these characteristics and molecular genetic factors. Conducting this research will contribute to the elucidation and advancement of a multidisciplinary therapeutic-diagnostic pathway. The study will utilise surgical specimens, irrespective of the disease stage, that have been formalin-fixed and paraffin-embedded. These specimens were previously collected for clinical practise at the Ocular Oncology of Fondazione Policlinico A. Gemelli IRCCS The informed consent of the patients regarding the use of these specimens for research purposes was obtained beforehand.Each specimen will be subjected to a comprehensive microscopic examination, followed by precise subclassification in accordance with the WHO classification and immunophenotypic characterization. An exhaustive collection of conventionally standardised histopathological prognostic attributes for sebaceous carcinomas will be compiled. Following this, tissue samples are sent for single and/or multiple IHC. Tumour tissues will be subjected to automated digital quantification in conjunction with multiparametric cell line evaluation. Integrating IHC with digital automation of analysis.Exome sequencing will be performed on DNA extracted from paraffin-embedded sections in order to detect variants that are specific to tumours.

For each tumour, three to nine sections (10 micrometres in thickness) will be utilised as the DNA source. Following the identification and separation of tumour tissue from normal tissue by the pathologist, the two DNAs will be sequenced independently. A comparison will be made between variants derived from tumour and normal tissue, with contrasting results. Anticipated outcomes include 1) somatic or tumor-specific variants, which are non-existent in healthy tissue, and 2) variants that are lost during the evolution of the tumour as a result of segmental chromosomal deletion or other mechanisms that induce heterozygosity loss. During the project's prospective phase, newly developed tumours will be preserved. Furthermore, this resource will facilitate methylome analysis, which is in addition to exome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Diagnosis of sebaceous Ca of the ocular adnexa
* Ability to obtain formalin-fixed and paraffin-embedded primary and/or metastatic tumour tissue (FFPE) and healthy tissue
* Availability of primary and/or metastatic tumour tissue in paraffin-embedded or OCT (prospective part) and healthy tissue
* Written informed consent for use of data for research purposes.

Exclusion Criteria:

* Age < 18 years;
* Lack of sufficient clinical data on selected patients.
* Lack of tumor and/or metastatic tissue in kerosene or OCT.
* Refusal to give informed consent to data processing for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-10-06 (Estimated); Study Completion 2025-10-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of different molecules in Microscopic and immunophenotypic analysis | 1 year
  Tissue samples will then be sent for single and/or multiple immunohistochemistry.

SECONDARY OUTCOMES:
Rate of somatic variants, variants with loss of heterozygosity, global mutational signature and identification of probable driver mutations | 1 year
  Rate of somatic variants, variants with loss of heterozygosity, global mutational signature and identification of probable driver mutations by exome sequencing;
Rate of correlations histopathological features with tumour DNA variants and disease stage. | 2 years
  Rate of correlations between histopathological features with tumour DNA variants and disease stage.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavo Savino, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prieto-Granada C, Rodriguez-Waitkus P. Sebaceous Carcinoma of the Eyelid. Cancer Control. 2016 Apr;23(2):126-32. doi: 10.1177/107327481602300206. PMID 27218789
- [Background] Owen JL, Kibbi N, Worley B, Kelm RC, Wang JV, Barker CA, Behshad R, Bichakjian CK, Bolotin D, Bordeaux JS, Bradshaw SH, Cartee TV, Chandra S, Cho NL, Choi JN, Council ML, Demirci H, Eisen DB, Esmaeli B, Golda N, Huang CC, Ibrahim SF, Jiang SB, Kim J, Kuzel TM, Lai SY, Lawrence N, Lee EH, Leitenberger JJ, Maher IA, Mann MW, Minkis K, Mittal BB, Nehal KS, Neuhaus IM, Ozog DM, Petersen B, Rotemberg V, Samant S, Samie FH, Servaes S, Shields CL, Shin TM, Sobanko JF, Somani AK, Stebbins WG, Thomas JR, Thomas VD, Tse DT, Waldman AH, Wong MK, Xu YG, Yu SS, Zeitouni NC, Ramsay T, Reynolds KA, Poon E, Alam M. Sebaceous carcinoma: evidence-based clinical practice guidelines. Lancet Oncol. 2019 Dec;20(12):e699-e714. doi: 10.1016/S1470-2045(19)30673-4. PMID 31797796
- [Background] Alfaar AS, Suckert CN, Rehak M, Girbardt C. The epidemiology of adults' eyelid malignancies in Germany between 2009 and 2015; An analysis of 42,710 patients' data. Eur J Ophthalmol. 2022 Nov 4;33(2):11206721221125018. doi: 10.1177/11206721221125018. Online ahead of print. PMID 36330713
- [Background] Tryggvason G, Bayon R, Pagedar NA. Epidemiology of sebaceous carcinoma of the head and neck: implications for lymph node management. Head Neck. 2012 Dec;34(12):1765-8. doi: 10.1002/hed.22009. Epub 2012 Jan 20. PMID 22267270
- [Background] Gauthier AS, Campolmi N, Tumahai P, Kantelip B, Delbosc B. Sebaceous carcinoma of the eyelid and Muir-Torre syndrome. JAMA Ophthalmol. 2014 Aug;132(8):1025-8. doi: 10.1001/jamaophthalmol.2014.1026. No abstract available. PMID 24969841
- [Background] Ferreira I, Wiedemeyer K, Demetter P, Adams DJ, Arends MJ, Brenn T. Update on the pathology, genetics and somatic landscape of sebaceous tumours. Histopathology. 2020 Apr;76(5):640-649. doi: 10.1111/his.14044. Epub 2020 Mar 17. PMID 31821583
- [Background] Jagan L, Zoroquiain P, Bravo-Filho V, Logan P, Qutub M, Burnier MN Jr. Sebaceous adenomas of the eyelid and Muir-Torre Syndrome. Br J Ophthalmol. 2015 Jul;99(7):909-13. doi: 10.1136/bjophthalmol-2014-305873. Epub 2015 Jan 16. PMID 25595178
- [Background] Yeatts RP, Waller RR. Sebaceous carcinoma of the eyelid: pitfalls in diagnosis. Ophthalmic Plast Reconstr Surg. 1985;1(1):35-42. doi: 10.1097/00002341-198501000-00006. PMID 3940100
- [Background] Orr CK, Yazdanie F, Shinder R. Current review of sebaceous cell carcinoma. Curr Opin Ophthalmol. 2018 Sep;29(5):445-450. doi: 10.1097/ICU.0000000000000505. PMID 29985175
- [Background] Kumar T, Tewari P, Khanna N, Surabhi, Bharti S, Sinha R, Bhadani PP. Cytomorphology of sebaceous carcinoma of the eyelid: A short series of three cases with literature review. Diagn Cytopathol. 2022 Dec;50(12):E361-E366. doi: 10.1002/dc.25029. Epub 2022 Aug 6. PMID 35932255
- [Background] Tetzlaff MT, Curry JL, Ning J, Sagiv O, Kandl TL, Peng B, Bell D, Routbort M, Hudgens CW, Ivan D, Kim TB, Chen K, Eterovic AK, Shaw K, Prieto VG, Yemelyanova A, Esmaeli B. Distinct Biological Types of Ocular Adnexal Sebaceous Carcinoma: HPV-Driven and Virus-Negative Tumors Arise through Nonoverlapping Molecular-Genetic Alterations. Clin Cancer Res. 2019 Feb 15;25(4):1280-1290. doi: 10.1158/1078-0432.CCR-18-1688. Epub 2018 Nov 12. PMID 30420449
- [Background] McGrath LA, Currie ZI, Mudhar HS, Tan JHY, Salvi SM. Management of recurrent sebaceous gland carcinoma. Eye (Lond). 2020 Sep;34(9):1685-1692. doi: 10.1038/s41433-019-0756-9. Epub 2020 Jan 2. PMID 31896805
- [Background] Magazin M, Dalvin LA, Salomao DR, Castner NB, Halbach C, Tooley AA. Sebaceous Carcinoma of the Eyelid: Proposed Nomenclature for Multifocal and Multicentric Disease. Ophthalmic Plast Reconstr Surg. 2023 Mar-Apr 01;39(2):117-122. doi: 10.1097/IOP.0000000000002281. Epub 2022 Oct 20. PMID 36356187